CLINICAL TRIAL: NCT00230152
Title: Nuclear Medicine for the Evaluation of Infection-the Added Value of Hybrid Imaging Modalities
Brief Title: Hybrid Imaging Modalities for the Evaluation of Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Rambam Health Care Campus, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: infectionCTIL
Record Dates: First submitted 2005-09-29; First posted 2005-09-30 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2005-09

CONDITIONS: Infectious Diseases
MeSH Terms: conditions — Communicable Diseases | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Imaging

SUMMARY:
The synergistic value of the fusion of physiologic and anatomical data has been described using several co-registration techniques for various nuclear medicine procedures and morphologic imaging modalities (single photon emission computed tomography-computed tomography [SPECT-CT], SPECT-magnetic resonance imaging [MRI], camera-based positron emission tomography [PET]-CT and PET-CT). The researchers hypothesize that fusion of nuclear medicine (NM) and CT data acquired sequentially in a single imaging session on one device is clinically superior to side-by-side evaluation of separately performed imaging tests. They hypothesize that more accurate localization of increased radiotracer activity on NM procedures will improve the diagnostic accuracy for detection of infection and will subsequently have a significant impact on patient management.

The purpose of the present study is to assess the clinical value of this new technology of fused imaging in patients undergoing diagnostic nuclear medicine evaluation for suspicion of an infection process.

DETAILED DESCRIPTION:
The researchers hypothesize that fusion of nuclear medicine (NM) and CT data acquired sequentially in a single imaging session on one device is clinically superior to side-by-side evaluation of separately performed imaging tests. They hypothesize that more accurate localization of increased radiotracer activity on NM procedures will improve the diagnostic accuracy for detection of infection and will subsequently have a significant impact on patient management.

The purpose of the present study is to assess the clinical value of this new technology of fused imaging in patients undergoing diagnostic nuclear medicine evaluation for suspicion of an infection process.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for NM imaging procedures to assess the presence of infectious processes.
* Patients signed informed consent

Exclusion Criteria:

* The study will not be performed in pregnant or lactating women.
* Patients unable or unwilling to tolerate the scan until its completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-02; Primary Completion 2007-04 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The impact of the imaging modality on patient management | 3 years

SECONDARY OUTCOMES:
The impact of the imaging modality on patient management | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Keidar, MD, PhD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel